CLINICAL TRIAL: NCT05769192
Title: Investigation of the Effects of Classical Massage Application on Individuals With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/03/04
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will be applied classical physiotherapy and classical massage
  Interventions: Other: Classical physiotherapy and classical massage
- Group 2 (Placebo Comparator): Group 2 will be applied classical physiotherapy and placebo massage
  Interventions: Other: Classical physiotherapy and placebo massage

INTERVENTIONS:
Other: Classical physiotherapy and classical massage — Within the scope of classical physiotherapy, hot pack will be applied for 20 minutes to the muscles in the lumbar region in the prone position. Stretching and strengthening exercises for the abdominal, lumbar and hip muscles will be given. Classical massage, known as Swedish massage, will be applied on the lumbar region in prone position. All applications will be done 5 days a week for 3 weeks.
  Arms: Group 1
Other: Classical physiotherapy and placebo massage — Within the scope of classical physiotherapy, hot pack will be applied for 20 minutes to the muscles in the lumbar region in the prone position. Stretching and strengthening exercises for the abdominal, lumbar and hip muscles will be given. In addition, placebo massage, applied without using any technique, will be applied to the lumbar region in the prone position. All applications will be done 5 days a week for 3 weeks.
  Arms: Group 2

SUMMARY:
The aim of this study is to examine the effects of classical massage on pain, spinal mobility, functional and psychological state, and life quality in individuals with chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is one of the most common problems in society, experienced by 70-80% of individuals at least once in their lifetime. Physical pain can cause serious functional losses that affect independence in daily life. In patients with low back pain, physical endurance decreases because of pain, spasm, decrease in muscle strength and deteriorated posture, and the functional capacity and quality of life of the patient are negatively affected. While most individuals recover spontaneously, 2-8% of them require medical treatment, and the response to conservative treatment is generally good. Along with medical treatment, different physiotherapy methods (electro-physical agents, massage, traction, exercises, etc.), which are conservative treatment methods, are also frequently used. It is known that classical physiotherapy modalities (heating agents and exercise approaches) have an important place in the treatment of these patients due to their positive effects on pain, strength, flexibility and functionality. Massage is used to systematically manipulate the soft tissues of the body with rhythmic pressure and to provide or maintain health. Basically, massage is a simple way to provide pain relief through physical and mental relaxation. It is thought to relieve pain in various ways, including increasing the pain threshold by secreting endorphins and closing the pain gate at the spinal cord level. Classical massage is considered rehabilitative and is also used to reduce symptoms associated with medical conditions. It has been reported that classical massage reduces many physical and psychological symptoms in different musculoskeletal problems (neck pain, fibromyalgia, etc.). However, there is a need for placebo-controlled studies in the literature examining the effects of classical massage in individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* Having non-specific low back pain lasting at least 3 months,
* Individuals willing to participate in the study

Exclusion Criteria:

* Having different pain syndromes (eg fibromyalgia)
* Having a history of spinal surgery or invasive examination in the last 6 months,
* Having a neurological or psychiatric disease
* Any ongoing related pathology (eg spondylolisthesis, fractures, tumor, osteoporosis or infection),
* Those with pregnancy status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | change from baseline at 3 weeks
  Pain intensity will be evaluated with a 10 cm Visual Analog Scale (VAS). The VAS is scored on a 10 cm horizontal line, with 0 meaning "no pain" and 10 "worst pain imaginable". Patients will be asked to mark their lower back pain on the horizontal line.

SECONDARY OUTCOMES:
Spinal mobility | change from baseline at 3 weeks
  Spinal mobility will be assessed with the Modified Shober test. With the patient in an upright position, a mark will be made at the midpoint of the imaginary line joining the posterior superior iliac spine on the back. Another mark will be made 10 cm above and 5 cm below this mark. The patient will be asked to lean forward maximally, keeping the knees fully extended. The distance between these marks will be measured. Mobility will be recorded by calculating the difference between the upright and maximum flexion end positions. It is stated that the greater the difference, the greater the mobility.
Functional status | change from baseline at 3 weeks
  Functional status will be assessed with the Oswestry Disability Index (ODI) . The index consists of 10 items (pain severity, personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life, travel) and is scored on a 0-5-point scale based on functional performance. Higher scores indicate more severe disability.
Psychological state | change from baseline at 3 weeks
  Psychological state will be evaluated using the Hospital Anxiety Depression Scale. The scale has 14 items, 7 of which with odd numbers represent anxiety while the other 7 with even numbers represent depression.
  Higher scores indicate more severe anxiety or depression.
Life quality | change from baseline at 3 weeks
  Life quality will be evaluated with the Short Form (SF-36) consisting of 36 items. It includes eight different fields: general health, bodily pain, physical function, physical and mental role limitations, mental health, vitality, and social function. The eight fields can be join mainly the physical component summary and the mental component summary that reflects physical and mental health. While '100' is the best score the '0' is the worst and higher scores indicate better life quality.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University